CLINICAL TRIAL: NCT05717660
Title: APalutamide and stEReotactic Body Radiation Therapy for Low Burden Metastatic Hormone senSItive Prostate Cancer, a rANdomized Trial - PERSIAN
Brief Title: APalutamiAPalutamide and stEReotactic Body Radiation Therapy for Metastatic Prostate Cancer
Acronym: PERSIAN
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Principal Investigator, Lorenzo Livi, Full Professor, Azienda Ospedaliero-Universitaria Careggi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PERSIAN
Record Dates: First submitted 2023-01-20; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Oligometastatic Hormone Sensitive Prostate Cancer

STUDY DESIGN:
Intervention Model Description: Patients will be randomized between control arm (Androgen Deprivation therapy and Apalutamide) or treatment arm (Androgen Deprivation therapy and Apalutamide and SBRT on all sites of metastatic disease)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Active Comparator): Androgen Deprivation therapy and Apalutamide
  Interventions: Combination Product: SBRT on all sites of metastatic disease+Apalutamide
- Treatment (Experimental): Androgen Deprivation therapy and Apalutamide and SBRT on all sites of metastatic disease
  Interventions: Combination Product: SBRT on all sites of metastatic disease+Apalutamide

INTERVENTIONS:
Combination Product: SBRT on all sites of metastatic disease+Apalutamide — oral Apalutamide 240 mg daily+ stereotactic body radiotherapy on all metastatic sites of disease, administered in 1-8 fractions for a total EQD2 of 50 Gy with an alpha/beta of 10.

SUMMARY:
Final results from TITAN trial showed that apalutamide plus ADT improved OS in a population of patients with metastatic hormone sensitive prostate cancer (mHSPC), if compared to ADT alone. However, stereotactic body radiotherapy (SBRT) showed to improve outcomes of oligometastatic patients if compared to systemic therapy alone within modern randomized trial, including a mixed cohort of different pathologies. However, there are no trials specifically exploring the benefit offered by SBRT in oligometastatic mHSPC treated with Apalutamide if compared to Apalutamide alone associated to Androgen deprivation therapy. Thus, a randomized trial was designed to test specifically the hypotesis that SBRT will improve outcome in a selected population of oligometastatic mHSPC treated with Apalutamide and ADT, undergoing baseline staging according to local reimbursability.

DETAILED DESCRIPTION:
Prospective Phase II randomized superiority study, open label, multicentric. Patients with Oligometastatic hormone sensitive prostate cancer defined as presence of ≤ 5 non-visceral metastatic lesions and treated with androgen deprivation treatment associated with Apalutamide will be randomized to receive standard systemic treatment alone or concomitant SBRT on all sites of metastatic disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have signed written informed consent
* Adult patients ≥ 18 years
* Oligometastatic hormone sensitive prostate cancer defined as presence of ≤ 5 non-visceral metastatic lesions *, **
* All lesions must be amenable to SBRT in judgment of treating radiation oncologist ***
* Patients with metastatic recurrence after previous radical prostatectomy or definitive radiotherapy will be included in the trial, provided that radical approach on prostate is administered
* Androgen deprivation therapy (ADT) started ≤ 6 months before enrollment
* Patients should be eligible to Apalutamide treatment

Exclusion Criteria:

* Presence of visceral disease
* De novo metastatic disease
* Any contraindication to the use of Apalutamide
* Any condition for which, in the opinion of the treating physician, SBRT should not be proposed or could be contraindicated

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-03-11 (Estimated); Primary Completion 2024-09-11 (Estimated); Study Completion 2025-03-11 (Estimated)

PRIMARY OUTCOMES:
Complete biochemical response | 6 months after treatment start.
  Rate of patients with complete biochemical response (PSA < 0.2 ng/ml)

SECONDARY OUTCOMES:
Freedom from biochemical progression | 2 years after treatment
  Biochemical progression defined according to Prostate Cancer Working Group Criteria
Freedom from radiological progression | 2 years after treatment
  radiological progression defined according to Prostate Cancer Working Group Criteria
Rate of adverse events | 2 years after treatment
  measured according to Common Terminology Criteria for Adverse Events
Overall Survival | 2 years after treatment
  Time between randomization and death from any cause
Cancer Specific Survival | 2 years after treatment
  Time between randomization and death from prostate cancer
Health related quality of life | 2 years after treatment
  Measured with European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30 questionnaire.
Health related quality of life | 2 years after treatment
  Measured with EORTC QLQ-PR25 questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- AOU Careggi Radiation Oncology Unit, Florence, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Palma DA, Olson R, Harrow S, Gaede S, Louie AV, Haasbeek C, Mulroy L, Lock M, Rodrigues GB, Yaremko BP, Schellenberg D, Ahmad B, Senthi S, Swaminath A, Kopek N, Liu M, Moore K, Currie S, Schlijper R, Bauman GS, Laba J, Qu XM, Warner A, Senan S. Stereotactic Ablative Radiotherapy for the Comprehensive Treatment of Oligometastatic Cancers: Long-Term Results of the SABR-COMET Phase II Randomized Trial. J Clin Oncol. 2020 Sep 1;38(25):2830-2838. doi: 10.1200/JCO.20.00818. Epub 2020 Jun 2. PMID 32484754
- [Background] Sweeney C, Bracarda S, Sternberg CN, Chi KN, Olmos D, Sandhu S, Massard C, Matsubara N, Alekseev B, Parnis F, Atduev V, Buchschacher GL Jr, Gafanov R, Corrales L, Borre M, Stroyakovskiy D, Alves GV, Bournakis E, Puente J, Harle-Yge ML, Gallo J, Chen G, Hanover J, Wongchenko MJ, Garcia J, de Bono JS. Ipatasertib plus abiraterone and prednisolone in metastatic castration-resistant prostate cancer (IPATential150): a multicentre, randomised, double-blind, phase 3 trial. Lancet. 2021 Jul 10;398(10295):131-142. doi: 10.1016/S0140-6736(21)00580-8. PMID 34246347
- [Background] Saad F, Chi KN, Shore ND, Graff JN, Posadas EM, Lattouf JB, Espina BM, Zhu E, Yu A, Hazra A, De Meulder M, Mamidi RNVS, Bradic B, Francis P, Hayreh V, Rezazadeh Kalebasty A. Niraparib with androgen receptor-axis-targeted therapy in patients with metastatic castration-resistant prostate cancer: safety and pharmacokinetic results from a phase 1b study (BEDIVERE). Cancer Chemother Pharmacol. 2021 Jul;88(1):25-37. doi: 10.1007/s00280-021-04249-7. Epub 2021 Mar 22. PMID 33754187
- [Background] Nuhn P, De Bono JS, Fizazi K, Freedland SJ, Grilli M, Kantoff PW, Sonpavde G, Sternberg CN, Yegnasubramanian S, Antonarakis ES. Update on Systemic Prostate Cancer Therapies: Management of Metastatic Castration-resistant Prostate Cancer in the Era of Precision Oncology. Eur Urol. 2019 Jan;75(1):88-99. doi: 10.1016/j.eururo.2018.03.028. Epub 2018 Apr 16. PMID 29673712
- [Background] Hellman S, Weichselbaum RR. Oligometastases. J Clin Oncol. 1995 Jan;13(1):8-10. doi: 10.1200/JCO.1995.13.1.8. No abstract available. PMID 7799047
- [Background] Phillips R, Shi WY, Deek M, Radwan N, Lim SJ, Antonarakis ES, Rowe SP, Ross AE, Gorin MA, Deville C, Greco SC, Wang H, Denmeade SR, Paller CJ, Dipasquale S, DeWeese TL, Song DY, Wang H, Carducci MA, Pienta KJ, Pomper MG, Dicker AP, Eisenberger MA, Alizadeh AA, Diehn M, Tran PT. Outcomes of Observation vs Stereotactic Ablative Radiation for Oligometastatic Prostate Cancer: The ORIOLE Phase 2 Randomized Clinical Trial. JAMA Oncol. 2020 May 1;6(5):650-659. doi: 10.1001/jamaoncol.2020.0147. PMID 32215577
- [Background] Ost P, Reynders D, Decaestecker K, Fonteyne V, Lumen N, De Bruycker A, Lambert B, Delrue L, Bultijnck R, Claeys T, Goetghebeur E, Villeirs G, De Man K, Ameye F, Billiet I, Joniau S, Vanhaverbeke F, De Meerleer G. Surveillance or Metastasis-Directed Therapy for Oligometastatic Prostate Cancer Recurrence: A Prospective, Randomized, Multicenter Phase II Trial. J Clin Oncol. 2018 Feb 10;36(5):446-453. doi: 10.1200/JCO.2017.75.4853. Epub 2017 Dec 14. PMID 29240541
- [Background] Zilli T, Achard V, Dal Pra A, Schmidt-Hegemann N, Jereczek-Fossa BA, Lancia A, Ingrosso G, Alongi F, Aluwini S, Arcangeli S, Blanchard P, Conde Moreno A, Counago F, Crehange G, Dirix P, Gomez Iturriaga A, Guckenberger M, Pasquier D, Sargos P, Scorsetti M, Supiot S, Tree AC, Zapatero A, Le Guevelou J, Ost P, Belka C. Recommendations for radiation therapy in oligometastatic prostate cancer: An ESTRO-ACROP Delphi consensus. Radiother Oncol. 2022 Nov;176:199-207. doi: 10.1016/j.radonc.2022.10.005. Epub 2022 Oct 10. PMID 36228761
- [Background] Bolla M, Collette L, Blank L, Warde P, Dubois JB, Mirimanoff RO, Storme G, Bernier J, Kuten A, Sternberg C, Mattelaer J, Lopez Torecilla J, Pfeffer JR, Lino Cutajar C, Zurlo A, Pierart M. Long-term results with immediate androgen suppression and external irradiation in patients with locally advanced prostate cancer (an EORTC study): a phase III randomised trial. Lancet. 2002 Jul 13;360(9327):103-6. doi: 10.1016/s0140-6736(02)09408-4. PMID 12126818
- [Background] Bolla M, Van Tienhoven G, Warde P, Dubois JB, Mirimanoff RO, Storme G, Bernier J, Kuten A, Sternberg C, Billiet I, Torecilla JL, Pfeffer R, Cutajar CL, Van der Kwast T, Collette L. External irradiation with or without long-term androgen suppression for prostate cancer with high metastatic risk: 10-year results of an EORTC randomised study. Lancet Oncol. 2010 Nov;11(11):1066-73. doi: 10.1016/S1470-2045(10)70223-0. Epub 2010 Oct 7. PMID 20933466
- [Background] Denham JW, Steigler A, Lamb DS, Joseph D, Turner S, Matthews J, Atkinson C, North J, Christie D, Spry NA, Tai KH, Wynne C, D'Este C. Short-term neoadjuvant androgen deprivation and radiotherapy for locally advanced prostate cancer: 10-year data from the TROG 96.01 randomised trial. Lancet Oncol. 2011 May;12(5):451-9. doi: 10.1016/S1470-2045(11)70063-8. PMID 21440505
- [Background] Horwitz EM, Bae K, Hanks GE, Porter A, Grignon DJ, Brereton HD, Venkatesan V, Lawton CA, Rosenthal SA, Sandler HM, Shipley WU. Ten-year follow-up of radiation therapy oncology group protocol 92-02: a phase III trial of the duration of elective androgen deprivation in locally advanced prostate cancer. J Clin Oncol. 2008 May 20;26(15):2497-504. doi: 10.1200/JCO.2007.14.9021. Epub 2008 Apr 14. PMID 18413638
- [Background] Goodwin JF, Schiewer MJ, Dean JL, Schrecengost RS, de Leeuw R, Han S, Ma T, Den RB, Dicker AP, Feng FY, Knudsen KE. A hormone-DNA repair circuit governs the response to genotoxic insult. Cancer Discov. 2013 Nov;3(11):1254-71. doi: 10.1158/2159-8290.CD-13-0108. Epub 2013 Sep 11. PMID 24027197
- [Background] Pilepich MV, Winter K, Lawton CA, Krisch RE, Wolkov HB, Movsas B, Hug EB, Asbell SO, Grignon D. Androgen suppression adjuvant to definitive radiotherapy in prostate carcinoma--long-term results of phase III RTOG 85-31. Int J Radiat Oncol Biol Phys. 2005 Apr 1;61(5):1285-90. doi: 10.1016/j.ijrobp.2004.08.047. PMID 15817329
- [Background] Warde P, Mason M, Ding K, Kirkbride P, Brundage M, Cowan R, Gospodarowicz M, Sanders K, Kostashuk E, Swanson G, Barber J, Hiltz A, Parmar MK, Sathya J, Anderson J, Hayter C, Hetherington J, Sydes MR, Parulekar W; NCIC CTG PR.3/MRC UK PR07 investigators. Combined androgen deprivation therapy and radiation therapy for locally advanced prostate cancer: a randomised, phase 3 trial. Lancet. 2011 Dec 17;378(9809):2104-11. doi: 10.1016/S0140-6736(11)61095-7. Epub 2011 Nov 2. PMID 22056152
- [Background] Widmark A, Klepp O, Solberg A, Damber JE, Angelsen A, Fransson P, Lund JA, Tasdemir I, Hoyer M, Wiklund F, Fossa SD; Scandinavian Prostate Cancer Group Study 7; Swedish Association for Urological Oncology 3. Endocrine treatment, with or without radiotherapy, in locally advanced prostate cancer (SPCG-7/SFUO-3): an open randomised phase III trial. Lancet. 2009 Jan 24;373(9660):301-8. doi: 10.1016/S0140-6736(08)61815-2. Epub 2008 Dec 16. PMID 19091394
- [Background] Smith MR, Saad F, Chowdhury S, Oudard S, Hadaschik BA, Graff JN, Olmos D, Mainwaring PN, Lee JY, Uemura H, Lopez-Gitlitz A, Trudel GC, Espina BM, Shu Y, Park YC, Rackoff WR, Yu MK, Small EJ; SPARTAN Investigators. Apalutamide Treatment and Metastasis-free Survival in Prostate Cancer. N Engl J Med. 2018 Apr 12;378(15):1408-1418. doi: 10.1056/NEJMoa1715546. Epub 2018 Feb 8. PMID 29420164
- [Background] Scher HI, Morris MJ, Stadler WM, Higano C, Basch E, Fizazi K, Antonarakis ES, Beer TM, Carducci MA, Chi KN, Corn PG, de Bono JS, Dreicer R, George DJ, Heath EI, Hussain M, Kelly WK, Liu G, Logothetis C, Nanus D, Stein MN, Rathkopf DE, Slovin SF, Ryan CJ, Sartor O, Small EJ, Smith MR, Sternberg CN, Taplin ME, Wilding G, Nelson PS, Schwartz LH, Halabi S, Kantoff PW, Armstrong AJ; Prostate Cancer Clinical Trials Working Group 3. Trial Design and Objectives for Castration-Resistant Prostate Cancer: Updated Recommendations From the Prostate Cancer Clinical Trials Working Group 3. J Clin Oncol. 2016 Apr 20;34(12):1402-18. doi: 10.1200/JCO.2015.64.2702. Epub 2016 Feb 22. PMID 26903579
- [Background] Chi KN, Agarwal N, Bjartell A, Chung BH, Pereira de Santana Gomes AJ, Given R, Juarez Soto A, Merseburger AS, Ozguroglu M, Uemura H, Ye D, Deprince K, Naini V, Li J, Cheng S, Yu MK, Zhang K, Larsen JS, McCarthy S, Chowdhury S; TITAN Investigators. Apalutamide for Metastatic, Castration-Sensitive Prostate Cancer. N Engl J Med. 2019 Jul 4;381(1):13-24. doi: 10.1056/NEJMoa1903307. Epub 2019 May 31. PMID 31150574
- [Background] Saad F, Cella D, Basch E, Hadaschik BA, Mainwaring PN, Oudard S, Graff JN, McQuarrie K, Li S, Hudgens S, Lawson J, Lopez-Gitlitz A, Yu MK, Smith MR, Small EJ. Effect of apalutamide on health-related quality of life in patients with non-metastatic castration-resistant prostate cancer: an analysis of the SPARTAN randomised, placebo-controlled, phase 3 trial. Lancet Oncol. 2018 Oct;19(10):1404-1416. doi: 10.1016/S1470-2045(18)30456-X. Epub 2018 Sep 10. PMID 30213449
- [Result] Chi KN, Chowdhury S, Bjartell A, Chung BH, Pereira de Santana Gomes AJ, Given R, Juarez A, Merseburger AS, Ozguroglu M, Uemura H, Ye D, Brookman-May S, Mundle SD, McCarthy SA, Larsen JS, Sun W, Bevans KB, Zhang K, Bandyopadhyay N, Agarwal N. Apalutamide in Patients With Metastatic Castration-Sensitive Prostate Cancer: Final Survival Analysis of the Randomized, Double-Blind, Phase III TITAN Study. J Clin Oncol. 2021 Jul 10;39(20):2294-2303. doi: 10.1200/JCO.20.03488. Epub 2021 Apr 29. PMID 33914595